CLINICAL TRIAL: NCT02659813
Title: ArchWire-RaCE: Orthodontic Archwires: a Randomised Clinical Trial of Effectiveness
Brief Title: Orthodontic Archwire Effectiveness Trial
Acronym: ArchWireRaCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Ormco Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015DE11
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Malocclusion
Keywords: Orthodontic wires
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Firewire (Experimental): Experimental Group 1. Novel orthodontic archwire.
  Interventions: Device: Orthodontic archwire
- CNiTi (Experimental): Experimental Group 2. Current best available orthodontic archwire
  Interventions: Device: Orthodontic archwire

INTERVENTIONS:
Device: Orthodontic archwire — Archwire used to align teeth in an orthodontic fixed brace
  Other Names: Firewire; Copper Nickel Titanium

SUMMARY:
This study protocol is for a randomised clinical trial which aims to test two materials used as orthodontic archwire to compare FireWire archwires to Copper Nickel Titanium (CNiTi) archwires. Both professional and patient related outcome measures are to be used to fully evaluate performance.

DETAILED DESCRIPTION:
This is a randomised clinical trial of Firewire and CNiTi as orthodontic aligning archwires. A two group single blind parallel multicentre study design in a National Health Service primary care setting in England will be used.

Patients will be recruited from those attending the practices for orthodontic treatment that meet the inclusion and exclusion criteria. Online randomisation will allocate to one of the two groups, stratified by centre and age group (adolescent / adult).

Sample size calculation indicates a total sample size of 42, but allowing for dropouts and missing data the investigators will recruit 64, 32 to each group.

Patients will be treated according to a strict clinical protocol including customised Damon Q fixed appliances and defined archwire sequence. Participants will be seen at initial 5 week intervals for data collection after new archwire placement, and otherwise at routine 10 week intervals.

Primary outcome data (rate of alignment) will be collected over the initial 10 weeks and secondary outcomes over the duration of the treatment (18 months approx).

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Class 1 Incisor relationship (British Standards Institute Classification)
* Labial segment crowding in upper and / or lower arch >4mm
* Little's Irregularity Index in upper and / or lower arch >4mm
* Eligible for NHS orthodontic treatment
* Planned non-extraction upper and lower fixed appliance orthodontic treatment

Exclusion Criteria:

* Previous fixed appliance orthodontic treatment
* Previous functional appliance treatment
* Planned use of fixed auxiliary appliances (e.g. quadhelix, Trans Palatal Arch)
* Cleft lip and palate or other craniofacial anomalies
* Hypodontia (excluding third molars), or missing teeth due to previous extraction
* Abnormal root morphology on pre-treatment radiographs
* Confirmed history of nickel allergy
* A medical history resulting in them taking analgesics for a chronic condition
* Limited mouth opening or other contra-indication to intra-oral scanning

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Rate of tooth movement | Initial six months of treatment
  Rate teeth move in response to force from archwire measured in millimetres on digital dental models

SECONDARY OUTCOMES:
Pain assessed by Visual Analogue Scale | Initial six months of treatment
  Visual Analogue Scale pain score after archwire placed
Tooth Root Resorption assessed on panoramic radiograph using method of Pandis et al (2008) | 18 months
  Damage to tooth root during tooth movement
Patient experience assessed by Questionnaire | Initial six months of treatment
  Questionnaire of patient experiences of braces

CONTACTS AND LOCATIONS:
Overall Officials: David R Bearn, BDS, PhD, Principal Investigator — University of Dundee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandis N, Nasika M, Polychronopoulou A, Eliades T. External apical root resorption in patients treated with conventional and self-ligating brackets. Am J Orthod Dentofacial Orthop. 2008 Nov;134(5):646-51. doi: 10.1016/j.ajodo.2007.01.032. PMID 18984396